CLINICAL TRIAL: NCT02893917
Title: A Randomized Phase 2 Study of Cediranib in Combination With Olaparib Versus Olaparib Alone in Men With Metastatic Castration Resistant Prostate Cancer
Brief Title: Testing Two Oral Drugs Combination (Cediranib and Olaparib) Compared to a Single Drug (Olaparib) for Men With Advanced Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01346; NCI-2016-01346 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000020461; 9984 (Other: Yale University Cancer Center LAO); 9984 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2016-09-08; First posted 2016-09-09 (Estimated); Results first posted 2025-03-30 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Advanced Prostate Adenocarcinoma With Neuroendocrine Differentiation; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma With Neuroendocrine Differentiation; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma With Neuroendocrine Differentiation; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cediranib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (olaparib, cediranib) (Experimental): Patients receive olaparib PO BID and cediranib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib; Drug: Olaparib
- Arm B (olaparib) (Active Comparator): Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Cediranib — Given PO
  Other Names: AZ-D2171; AZD 2171; AZD2171
  Arms: Arm A (olaparib, cediranib)
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This randomized phase II trial studies how well olaparib with or without cediranib works in treating patients with castration-resistant prostate cancer that has spread to other places in the body (metastatic). PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Cediranib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving olaparib and cediranib may help treat patients with castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the clinical activity of the combination of cediranib and olaparib, as measured by radiographic progression free survival (rPFS), as compared to olaparib monotherapy in patients with metastatic castration resistant prostate cancer (mCRPC).

SECONDARY OBJECTIVES:

I. To assess the clinical activity of the combination of cediranib and olaparib, as measured by prostate-specific antigen (PSA) response rate, radiographic response rate by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1, and overall survival (OS), as compared to olaparib monotherapy in patients with mCRPC.

II. To evaluate association of homologous recombination deoxyribonucleic acid (DNA) repair deficiency (HRD) with the clinical activity of the combination of cediranib and olaparib or olaparib monotherapy, as measured by rPFS, in mCRPC patients.

III. To evaluate the safety the combination of cediranib and olaparib and olaparib monotherapy in patients with metastatic prostate cancer.

EXPLORATORY OBJECTIVES:

I. To characterize genomic alterations by whole exome sequencing in mCRPC patients and correlate that with clinical activity or resistance to olaparib with or without cediranib.

II. To characterize changes in ribonucleic acid (RNA) expression of DNA repair genes, angiogenesis markers, and immune markers, by whole transcriptome sequencing and correlate with clinical activity or resistance to olaparib with or without cediranib.

III. To characterize changes in immune tumor microenvironment in mCRPC patients by profiling expression of co-stimulatory and co-inhibitory molecules and tumor infiltrating lymphocytes, and correlate with clinical activity or resistance to olaparib with or without cediranib.

IV. To identify baseline predictive biomarkers for rPFS or response and to identify on-treatment markers of acquired resistance in men with mCRPC receiving either olaparib plus cediranib or olaparib alone.

V. To explore biomarker signatures that correlate with the clinical activity or resistance to olaparib with or without cediranib, including changes in gene expression or acquired mutations in tumor biopsies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive olaparib orally (PO) twice daily (BID) and cediranib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive olaparib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed progressive, metastatic castration resistant prostate adenocarcinoma by meeting ALL the following:

  * Pathology of prostate gland or metastatic disease must confirm the diagnosis of prostate adenocarcinoma; mixed histology with other variants including but not limited to small cell or neuroendocrine differentiation must be discussed with the study principal investigator (PI)
  * Metastasis must be documented by radiographic evidence
  * Castration resistance must be documented with surgical or medical castration with serum testosterone < 50 ng/dL (< 2.0 nM); if the patient is being treated with luteinizing hormone-releasing hormone (LHRH) agonists (patient who has not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to cycle 1, day 1 and must be continued throughout the study
  * Progression must be evidenced and documented by any of the following parameters

    * Two consecutively rising PSA values, above the baseline, at a minimum of 1-week intervals; the minimal value to enter the study is 1.0 ng/ml or greater; the reference value (#1) is the last PSA measured before increases are documented, with subsequent values obtained a minimum of 1 week apart; if the PSA at time point 3 (value #3A) is greater than that at point 2, then eligibility has been met; if the PSA is not greater than point 2 (value #3B), but value #4 is, the patient is eligible assuming that other criteria are met, if values 3A or #4 are 1 ng/mL or higher (Prostate Cancer Working Group 3)
    * Appearance of one or more new lesions on bone scan
    * Progressive disease by RECIST 1.1
* Must have a tumor lesion safely accessible for biopsy per the investigator's discretion; while a soft tissue metastasis is preferred for a biopsy, a bone metastasis is allowed for biopsy as long as enough cores can be obtained; a biopsied lesion cannot be used for target lesion for response assessment
* Must be agreeable to the mandatory research tumor biopsies (pre-treatment and on-treatment); tumor biopsies are mandatory at pre-treatment and at on-treatment; there is an optional biopsy at post-progression
* Must have received at least one prior line of therapy for mCRPC; a taxane chemotherapy administered for metastatic castration sensitive disease will not count, unless patient develops disease progression within 12 months from the last dose chemotherapy
* Must have a life expectancy greater than or equal to 16 weeks
* If patient is currently on prednisone or other corticosteroids for palliation, the dose must be less than or equal to 10 mg a day or its equivalent dose and it must have been started at least 4 weeks prior to cycle 1 day 1
* Patients must have measurable disease by RECIST v1.1, or evaluable disease with bone metastases demonstrated by Tc99 bone scan; patients with bone metastases only are allowed (NOTE: nodes >= 1.5 cm (not >= 2 cm) in the short axis are considered measurable, per The Prostate Cancer Working Group 3 [PCWG3])
* Toxicities of prior therapy (except alopecia) should be resolved to =< grade 1 as per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0; patients with long-standing stable grade 2 neuropathy or others (e.g., adrenal insufficiency or hypothyroidism on stable doses of replacement therapy) may be allowed after discussion with the study principal investigator (PI)
* Age >= 18 years. There is no dosing or adverse event data currently available on the use of cediranib or olaparib in patients < 18 years of age, thus excluding them from enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >= 70%)
* White blood count (WBC) > 3 x 10^9/L (within 28 days prior to administration of study treatment)
* Absolute neutrophil count >= 1,500/mcL (within 28 days prior to administration of study treatment)
* Platelets >= 100,000/mcL (within 28 days prior to administration of study treatment)
* Hemoglobin >= 10 g/dL with no pack red blood cell transfusion in the past 28 days (within 28 days prior to administration of study treatment)
* Creatinine clearance >= 51 mL/min, calculated using Cockcroft-Gault formula (within 28 days prior to administration of study treatment)
* Urine protein: creatinine ratio (UPC) of =< 1 (within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN) (within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) < 3 times institutional ULN unless liver metastases are present in which case they must be < 5 x ULN (within 28 days prior to administration of study treatment)
* Coagulation parameters (international normalized ratio [INR] and activated partial thromboplastin time [aPTT]) within 1.25 x ULN institutional limits, except where a lupus anti-coagulant has been confirmed, or except patients on anticoagulation (within 28 days prior to administration of study treatment)
* Patients must be able to swallow oral medications and not have gastrointestinal illnesses that would preclude absorption of cediranib or olaparib
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction; patients can be on thyroid hormone replacement medication; asymptomatic patients with elevated thyroid-stimulating hormone (TSH) with normal T4/T3 are allowed to enroll, and recommended to follow with routine thyroid function test especially if they are randomized to cediranib/olaparib arm
* Adequately controlled blood pressure (BP) < 140 mmHg (systolic) and < 90 mmHg (diastolic) taken in the clinic setting by a medical professional within 2 weeks prior to starting study; patients with hypertension may be managed with up to a maximum of 3 antihypertensive medications; patients who are on 3 antihypertensive medications are highly recommended to be followed by a cardiologist or blood pressure specialist for management of BP while on protocol
* Patients must be willing and able to check and record daily blood pressure readings when randomized to cediranib containing arm
* Patients must have documented left ventricular ejection fraction (LVEF) by echocardiogram greater than institution's lower limit of normal (or 55% if threshold for normal not otherwise specified by institutional guidelines) obtained within 3 months prior to registration if they have any of the following risk factors for cardiac toxicities:

  * A New York Heart Association (NYHA) classification of II controlled with treatment
  * Prior central thoracic radiation therapy (RT), including RT to the heart
  * History of myocardial infarction within 12 months prior to registration
  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab
  * Prior history of other significant impaired cardiac function
* Male participants and their female partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination (see below for acceptable methods), and not to donate sperm, throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner; acceptable methods of contraception to be used in this study include:

  * Condom with spermicide and one of the following:

    * Oral contraceptive or hormonal therapy (e.g. hormone implants)
    * Placement of an intra-uterine device
  * Acceptable non-hormonal birth control methods include:

    * Total sexual abstinence; abstinence must be for the total duration of the study and the drug washout period
    * Vasectomized sexual partner plus male condom; with participant assurance that partner received post-vasectomy confirmation of azoospermia
    * Tubal occlusion plus male condom with spermicide
    * Intrauterine device (IUD) plus male condom+spermicide; provided coils are copper-banded
  * Acceptable hormonal methods:

    * Etonogestrel implants (e.g., Implanon, Norplan) + male condom with spermicide
    * Normal and low dose combined oral pills + male condom with spermicide
    * Norelgestromin/ethinyl estradiol (EE) transdermal system + male condom with spermicide
    * Intravaginal device + male condom with spermicide (e.g., EE and etonogestrel)
    * Cerazette (desogestrel) + male condom with spermicide; cerazette is currently the only highly efficacious progesterone based pill
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, hormonal therapy (except LHRH agonist or antagonist), immunotherapy, radioisotope therapy, or RT within 21 days prior to start of the study agents
* Initiating bisphosphonate, or RANKL antibody therapy or adjusting the dose/regimen within 30 days prior to cycle 1 day 1 is prohibited; patients on a stable bisphosphonate regimen are eligible and may continue
* Patients who have received any other investigational agents within the past 28 days prior to cycle 1 day 1
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) scans are excluded from this clinical trial; while screening brain MRI is not required, it should be performed if clinically indicated at the discretion of the treating investigator; should patient found to have brain metastasis, treatment of brain metastasis must precede the participation in this study
* For patients with known and treated brain metastases is allowed in this study if they fulfill ALL of the following criteria:

  * The lesions have remained radiologically stable for at least six weeks after completion of brain irradiation or stereotactic brain radiosurgery, and must remain stable at the time of study entry
  * There is no mass effect present radiologically and no steroids requirement for symptom control for more than 4 weeks
* Patients who have received a prior inhibitor of vascular endothelial growth factor (VEGF) signaling inhibitor, or a poly adenosine diphosphate-ribose polymerase (PARP) inhibitor administered
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib or olaparib
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir), moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil), strong CYP3A inducers (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil); a minimum washout period of 2 weeks prior to cycle 1 day 1 is required for strong inhibitors, and at least one week for moderate inhibitors; a minimum washout period of 4 weeks prior to cycle 1 day 1 is required for CYP3A inducers; a minimum washout period of 5 weeks prior to cycle 1 day 1 is required for enzalutamide or phenobarbital; dihydropyridine calcium-channel blockers are permitted for management of hypertension
* Current use of natural herbal products or other "folk remedies"; if using previously, patients must stop using natural herbal products while participating in this study; multivitamin, calcium (Ca)/vitamin D (Vit D) and other vitamin complex supplements are allowed
* Patients with concomitant or prior invasive malignancies within the past 5 years; subjects with limited stage basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the breast, or non-muscle invasive bladder cancer, are eligible as long as they received curative intent therapy
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled seizures ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Resting ECG with corrected QT (QTc) > 470 msec on two or more time points within a 24 hour period, noted within 14 days of treatment, or family history of long QT syndrome
* History of myocardial infarction within 6 months of the randomization
* History of stroke or transient ischemic attack within 6 months of the randomization
* NYHA classification of III or IV
* Current cardiac arrhythmic condition requiring concurrent use of anti-arrhythmic drug; rate controlled atrial fibrillation is allows
* History of hypertensive crisis or hypertensive encephalopathy within 3 years of the randomization
* Clinically significant peripheral vascular disease or known abdominal aortic aneurysm ( > 5 cm in diameter) or history of aortic dissection; patients with known history of abdominal aortic aneurysm (AAA) with >= 4 cm in diameter, a repeat ultrasound (US) within the last 6 months prior to randomization will be required to document that it is =< 5 cm, and patient must be asymptomatic from the aneurysm, and the blood pressure must be well controlled as required in this protocol
* A major surgical procedure, open biopsy, or significant traumatic injury within 3 months prior to cycle 1 day 1 (percutaneous/endobronchial/endoscopic biopsies are allowed)
* History of bowel obstruction within 1 month prior to starting study drugs
* History of hemoptysis within the last 1 month prior to randomization
* Presence of cavitation of central pulmonary lesion, or radiographic evidence of pneumonitis or other extensive bilateral lung disease such as interstitial lung disease
* Any history of gastrointestinal (GI) perforation, history of intra-abdominal abscess within 3 months prior to starting treatment, or history of abdominal fistula unless the fistula history meets all the following: (a) the fistula was surgically repaired, (b) there has been no evidence of fistula for at least 6 months prior to starting treatment, (c) patient is deemed to be at low risk of recurrent fistula, and (d) the case must be discussed with the study PI
* Current dependency on intravenous (IV) hydration or total parenteral nutrition (TPN)
* Known coagulopathy or bleeding diathesis; those on therapeutic anticoagulation or anti-platelet agent are permitted only after discussing with the study PI
* Patients with history of intra-abdominal bleeding or retroperitoneal bleeding within the last 3 years are excluded
* Patients with myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML), or features suggestive of MDS/AML
* Patients with known active human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection; it is because of the potential requirement for anti-viral therapies that are prohibited on the study; patients with a history of hepatitis B or hepatitis C, who are deemed cured and no longer require treatment may be allowed to enroll after consultation with the respective specialist and the study PI
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment in the present study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2026-06-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Kim, Principal Investigator — Yale University Cancer Center LAO
Locations (16):
- United States (16):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Kim JW, McKay RR, Radke MR, Zhao S, Taplin ME, Davis NB, Monk P, Appleman LJ, Lara PN Jr, Vaishampayan UN, Zhang J, Paul AK, Bubley G, Van Allen EM, Unlu S, Huang Y, Loda M, Shapiro GI, Glazer PM, LoRusso PM, Ivy SP, Shyr Y, Swisher EM, Petrylak DP. Randomized Trial of Olaparib With or Without Cediranib for Metastatic Castration-Resistant Prostate Cancer: The Results From National Cancer Institute 9984. J Clin Oncol. 2023 Feb 1;41(4):871-880. doi: 10.1200/JCO.21.02947. Epub 2022 Oct 18. PMID 36256912

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Started | 45 | 45
Received Intervention | 44 | 45
Discontinued Treatment | 44 | 45
Completed (Included in the final analyses.) | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib) | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 81] | 70 [51 to 82] | 69 [48 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 45 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37 | 38 | 75
  Race: Non-White | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90
ECOG Performance Status Scale [Count of Participants; unit: Participants] — Count of participants where ECOG Performance Status Scale = 0 (Fully active, able to carry on all pre-disease performance without restriction)
  Participants | 22 | 23 | 45
Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 86.9 [0.30 to 3145] | 58.4 [0.02 to 1453] | 72.5 [0.02 to 3145]
Measurable disease (yes/no) [Count of Participants; unit: Participants]
  Yes | 31 | 33 | 64
  No | 14 | 12 | 26
Liver Metastases (Yes/No) [Count of Participants; unit: Participants]
  Yes | 10 | 10 | 20
  No | 35 | 35 | 70
Any Novel Hormonal Agent (Yes/No) [Count of Participants; unit: Participants] — Either in metastatic castration-sensitive prostate cancer or metastatic castration-resistant prostate cancer setting.
  Participants
    Yes | 45 | 43 | 88
    No | 0 | 2 | 2
Prior Cytotoxic Chemotherapy [Count of Participants; unit: Participants]
  1 cytotoxic chemotherapy | 17 | 20 | 37
  2 or more cytotoxic chemotherapies | 20 | 12 | 32
  no prior cytotoxic chemotherapy | 8 | 13 | 21

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival
Description: The two study arms will be compared for radiographic progression free survival with Kaplan-Meier estimates and log-rank tests. The Rothman confidence interval, which is based on Greenwood's variance, Thomas and Grunkemeier confidence interval, and the simultaneous confidence bands by Nair and Hall and Wellner, will be reported. In addition, the possible confounding variables will be compared for survival with log-rank test.
Time Frame: Time interval from random assignment to the date when the first site of disease is found to progress, or death, whichever occurs first, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 45 | 45
months | 8.5 [5.4 to 12.0] | 4.0 [3.2 to 8.5]
Statistical Analysis 1: Comparison: Arm A (Olaparib, Cediranib) vs Arm B (Olaparib); Test type: Superiority; p = 0.0359, Regression, Cox; Hazard Ratio (HR) = 0.617, 95% CI 2-sided [0.392 to 0.969]

2. Secondary Outcome: Overall Survival
Description: Will use the rank preserving structure failure time model for the overall survival analysis.
Time Frame: Time between randomization and death due to any cause (or last contact for surviving patients and those lost to follow-up), assessed up to 5 years
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 45 | 45
months | 11.8 [10.33 to NA] — Insufficient number of participants with events. | 17.3 [15.5 to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Arm A (Olaparib, Cediranib) vs Arm B (Olaparib); Test type: Superiority; Regression, Cox — no p value provided; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.705 to 2.399]

3. Secondary Outcome: Objective Response Rate
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1. The exact 95% confidence interval of objective response rate will be reported based on the binomial distribution. The multivariate data analysis will be completed using the logistic regression model. The adjusted p-value and adjusted 95% confidence interval will also be reported.
Time Frame: Up to 5 years
Population: 64 patients were evaluable for objective response by RECIST v1.1 criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 33 | 31
Participants | 6 | 4

4. Secondary Outcome: Prostate-specific Antigen Response Rate
Description: Prostate-specific antigen response will be defined by prostate-specific antigen decline from baseline > 50%, confirmed by a second value at 3-4 weeks later. Prostate-specific antigen response rate analysis will be based on a subset of patients who had prostate-specific antigen progression prior to enrollment. The multivariate data analysis will be completed using the logistic regression model.
Time Frame: Up to 5 years
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 45 | 45
Participants | 9 | 6

5. Secondary Outcome: Correlation Between Homologous Recombination Deficiency Status and Radiographic Progression Free Survival
Description: Homologous recombination deficiency positive status is defined by presence of homozygous deletion or deleterious mutations in key homologous recombination genes of deoxyribonucleic acid repair genes as analyzed by BROCA-homologous recombination test. The data analysis will be completed using log rank Test. The multivariate data analysis will be completed using the Cox PH model.
Time Frame: Up to 1 week prior to start of therapy
Population: Data are for those with evaluable data and then split by HRD status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 41 | 43
months
  HRD positive: number analyzed (Participants) | 12 | 14
  HRD positive | 10.63 [5.90 to NA] — Insufficient number of participants with events. | 3.83 [2.33 to NA] — Insufficient number of participants with events.
  HRD negative: number analyzed (Participants) | 29 | 29
  HRD negative | 5.47 [3.73 to 11.77] | 4.03 [3.73 to 8.47]
Statistical Analysis 1: Comparison: Arm A (Olaparib, Cediranib) vs Arm B (Olaparib); HRD positive ONLY; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.272 to 1.504]
Statistical Analysis 2: Comparison: Arm A (Olaparib, Cediranib) vs Arm B (Olaparib); HRD negative ONLY; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 0.777, 95% CI 2-sided [0.448 to 1.348]

6. Secondary Outcome: Incidence of Genomic Alterations
Description: Will be assessed by whole exome sequencing and transcriptome sequencing. The biomarker data analysis will be completed using Lasso-based elastic net method.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 45 | 45
Participants | 12 | 14

7. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (CTCAE version 5.0 will be effective by April 1, 2018). Descriptive statistics, including means, standard deviations, and ranges for continuous parameters, as well as percentages and frequencies for categorical parameters, will be presented. Adverse medical events will be tabulated. NCI toxicity grade 3 and grade 4 laboratory abnormalities will be listed and tabled. At the time of results reporting, presented are the count of participants in either arm that experienced at least 1 adverse event.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
Number analyzed (Participants) | 44 | 45
Participants | 44 | 45

8. Other Pre Specified Outcome: Baseline Predictive Biomarkers by Plasma Angiome
Description: The data analysis will be completed using Lasso-based elastic net method.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: On-treatment Markers of Acquired Resistance by Plasma Angiome
Description: The data analysis will be completed using Lasso-based elastic net method.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm A (Olaparib, Cediranib) | Arm B (Olaparib)
All-Cause Mortality (participants affected / at risk) | 35/44 | 34/45
Serious Adverse Events (participants affected / at risk) | 21/44 | 21/45
Other Adverse Events (participants affected / at risk) | 44/44 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Olaparib, Cediranib) (N=44) | Arm B (Olaparib) (N=45)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4
Anemia (Blood and lymphatic system disorders) | 3 | 4
Ascites (Gastrointestinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 3 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 4 | 0
Creatinine increased (Investigations) | 0 | 4
Death NOS (General disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3
Fatigue (General disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 0
Hematoma (Vascular disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Pain (General disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 2
Transient ischemic attacks (Nervous system disorders) | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Olaparib, Cediranib) (N=44) | Arm B (Olaparib) (N=45)
Fatigue (Nervous system disorders) | 29 | 23
Diarrhea (Gastrointestinal disorders) | 28 | 12
Anorexia (Metabolism and nutrition disorders) | 21 | 9
Hypertension (Endocrine disorders) | 20 | 0
Nausea (Gastrointestinal disorders) | 19 | 19
Anemia (Blood and lymphatic system disorders) | 14 | 19
Weight Loss (Metabolism and nutrition disorders) | 11 | 3
Vomiting (Gastrointestinal disorders) | 9 | 7
Hypothyroidism (Endocrine disorders) | 9 | 0
Plt count decreased (Investigations) | 8 | 7
WBC decreased (Investigations) | 7 | 6
Dysgeusia (Nervous system disorders) | 7 | 5
Constipation (Gastrointestinal disorders) | 6 | 4
Headache (Immune system disorders) | 6 | 4
Lymphocyte decreased (Investigations) | 6 | 7
Creatinine Increased (Investigations) | 4 | 5
Dizziness (Nervous system disorders) | 2 | 4
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT02893917/Prot_SAP_002.pdf
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT02893917/ICF_001.pdf